CLINICAL TRIAL: NCT00679484
Title: A 24-Week Multicentre, Randomized, Double-Blind, Controlled, Parallel Group Non-Inferiority Study to Assess the Efficacy and Safety of Olmesartan Medoxomil Versus Candesartan Cilexetil in Patients With Symptomatic Heart Failure (NYHA II-IV)
Brief Title: Study to Demonstrate the Non-inferiority of Olmesartan Medoxomil Versus Candesartan Cilexetil in Reducing Blood B-type (or Brain) Natriuretic Peptide Levels at Week 24
Acronym: OLMEBNP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of subject recruitment
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Senior Manager Clinical Development, Daiichi Sankyo Europe GmbH
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSE-866-45; 2007-003060-22 EUDRACT Number
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2010-08

CONDITIONS: Chronic Heart Failure; High Blood B-type (or Brain) Natriuretic Peptide (BNP) Level
MeSH Terms: interventions — Olmesartan Medoxomil; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: olmesartan medoxomil + candesartan cilexetil placebo
- 2 (Experimental)
  Interventions: Drug: olmesartan medoxomil placebo + candesartan cilexetil

INTERVENTIONS:
Drug: olmesartan medoxomil + candesartan cilexetil placebo — Dosage form: tablet; frequency: daily; duration: 24 weeks
  Arms: 1
Drug: olmesartan medoxomil placebo + candesartan cilexetil — Dosage form: tablets; frequency: daily; duration: 24 weeks
  Arms: 2

SUMMARY:
This study will compare olmesartan medoxomil to candesartan cilexetil in reducing BNP, a prognostic biomarker of heart failure, at week 24

ELIGIBILITY:
Inclusion Criteria:

* Male or female, adult, out-patients aged between 18 and 85 years
* Patients with documented hospital admission within the previous 3 months before randomization with discharge diagnosis of CHF
* Patients with functional NYHA class II-IV with LVEF < 40% assessed within the last 3 months
* Patients with blood BNP levels > 400 pg/ml or NT-ProBNP levels > 1500 pg/ml
* Patients with CHF due to ischemic heart disease, idiopathic dilated cardiomyopathy (IDC), mitral or aortic insufficiency or hypertension
* Patients with stable conventional treatment with diuretics, ACEI and/or beta-blockers and/or aldosterone antagonists for at least 2 months prior to randomisation, unless documented contraindication or intolerance

Exclusion Criteria:

* Females who are pregnant or plan a pregnancy during the time of the trial, are nursing or are of childbearing potential and not using acceptable methods of contraception. If a female becomes pregnant during the study, she has to be withdrawn immediately
* Patients with current hospitalisation due to heart failure
* Patients with stroke or transient ischemic attack (TIA) within the last 3 months
* Patients with acute coronary syndrome, myocardial infarction, coronary artery bypass or angioplasty within 3 months
* Planned cardiac surgery, revascularization or resynchronization within the study period
* Patients with operable valvular disease or significant obstructive cardiomyopathy
* Patients with bradycardia [heart rate (HR) < 50 bpm]
* Patients with hypotension [systolic blood pressure (SBP) < 90 mmHg]
* Patients with obstructive pneumopathy
* Patients with clinical significant renal failure (creatininemia > 200 micromol/l)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Absolute BNP change from week 0 to 24 of treatment | 24 weeks

SECONDARY OUTCOMES:
Proportion of BNP responders at week 4, 8, 16 and 24 (BNP levels reduced to 350 pg/ml or less at all time points) | 24 weeks maximum
BNP change from week 0 to week 4, 8, and 16 | 16 weeks maximum
Incidence of critical events at 24 weeks: All cause death; Cardiovascular death defined as death due to: HF, myocardial infarction, cardiac arrhythmia, stroke/cerebral vascular accident, other cardiovascular cause (e.g., aneurysm or pulmonary embolism) | 24 weeks
Event-free survival | 24 weeks
Time-to-death | 24 weeks
Time-to-first cardiovascular event | 24 weeks maximum
Change in clinical status: Improvement: patient alive without any cardiovascular event with an improvement of at least one NYHA functional class level; No change: patient alive without any cardiovascular event with stable functional NYHA class | 24 weeks

CONTACTS AND LOCATIONS:
Locations (11):
- France (7):
  - Bron
  - Cedex
  - Cholet
  - Langres
  - Mannheim
  - Pontoise
  - Roubaix
- Germany (3):
  - Bad Nauheim
  - Berlin
  - Lambrecht
- Ad Delft, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/